CLINICAL TRIAL: NCT01464515
Title: Feasibility Study in Order to Test the Efficiency of Deep TMS on Patient With MCI
Brief Title: Efficiency of Deep Transcranial Magnetic Stimulation on Patients With Mild Cognitive Impairment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: P-0021
Record Dates: First submitted 2011-10-25; First posted 2011-11-03 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment, So Stated; Deep Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real TMS (Active Comparator): this group will receive high frequency deep TMS treatment of 10HZ
  Interventions: Device: H-Coil Deep TMS
- SHAM TMS (Sham Comparator): this group will receive SHAM treatment of deep TMS
  Interventions: Device: SHAM Coil TMS

INTERVENTIONS:
Device: H-Coil Deep TMS — this group will receive high frequency treatment of deep TMS with 10Hz
  Arms: Real TMS
Device: SHAM Coil TMS — this group will receive SHAM treatment of deep TMS
  Arms: SHAM TMS

SUMMARY:
This is a first feasibility study in order to test if deep Transcranial Magnetic Stimulation (TMS) treatment with high frequency (10Hz) will improve the symptoms of patient MCI (Mild Cognitive impairment). The hypothesis of the study is that high frequency treatment with deep TMS will improve the daily functioning of patients who suffers from MCI.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 50-80 years of age.
2. Self reporting of the patient about memory deterioration, without any damage of daily lify functioning.
3. Scored of one standard deviation below the average (according to standardization of age and years of schooling) in the memory index and Mindstream test, without any major damage of other cognitive function)
4. score >= 24 in MMSE (Mini Mental State Examination) test.
5. Preserved Cognitive and executive functioning, without dementia according to DSM -IV
6. Lack of other reason for memory deterioration like acute affect disorder or other neurological disorders, according to the doctor diagnosis.
7. Score of maximum 0.5 in the Clinical Dementia Rating. in this test the score of the memory index will be 0.5 or 1, and not more then 1 point in two other index of this test.
8. Capable and willing to provide informed consent.

Exclusion Criteria:

1. Any other Axis I diagnosis as the primary diagnosis
2. Any medications that can cause a risk of seizure. for instance, anti psychotic medication, high dosage of anti depression medication
3. History of non tolerance for TMS treatment
4. Diagnosis of Severe personality disorder according to DSM-IV
5. current suicidal tendency
6. Uncontrolled hypertension
7. History of epilepsy, seizure, or heat convulsion
8. History of epilepsy or seizure in first degree relatives
9. History of head injury or stroke
10. History of metal implants in the head (except dental fillings)
11. History of surgery entailing metallic implants or known history of any metallic particles in the eye, implanted cardiac pacemaker, cochlear implants, use of neurostimulators, or any medical pumps
12. History of drug or alcohol abuse
13. Inadequate communication with examiner
14. Participation in another clinical study, either concurrent with this trial or in the 3 months preceding it
15. Inability to sign a consent form
16. Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Mindstreams | the test will be assessed on visit 17 which means 4 month from baseline
  Mindstreams test is designed to test the I.Q change of the patients from baseline

SECONDARY OUTCOMES:
CDR - Clinical Dementia Rating | the test will be assessed on visit 17 which means 4 month from baseline
  CDR test is designed to test the dementia severity of the patients from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Ash, Dr., Principal Investigator — Ichilov Hospital
Locations (1):
- Ichilov Hospital, Neurological Department, Tel Aviv, Israel